CLINICAL TRIAL: NCT00159107
Title: Acamprosate and Integrative Behavior Therapy in the Outpatient Treatment of Alcohol Dependents
Brief Title: Integrative Therapy in Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Addiction Research Network (Other); Merck Sharp & Dohme LLC (Industry); University of Bonn (Other); Universität Duisburg-Essen (Other); University of Homburg (Other); Psychosomatic Clinic of Bergisch Gladbach (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01EB0133
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2007-10

CONDITIONS: Alcoholism
Keywords: alcoholism; abstinence enhancement; psychotherapy; cognitive behavior therapy vs. supportive counseling; Acamprosate vs. Placebo; multi-center study
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): Placebo +Integrative behavior therapy
  Interventions: Behavioral: Integrative behavior therapy; Drug: Placebo
- 3 (Experimental): Acamprosate + treatment as usual
  Interventions: Drug: Acamprosate
- 1 (Experimental): Acamprosate + Integrative behavior therapy
  Interventions: Drug: Acamprosate; Behavioral: Integrative behavior therapy

INTERVENTIONS:
Drug: Acamprosate — Acamprosate
  Arms: 1; 3
Behavioral: Integrative behavior therapy — Integrative behavior therapy
  Arms: 1; 2
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The main aim of this project consists in the investigation of the interaction of behavior therapy and Acamprosate in the outpatient treatment of alcoholic patients in a randomized, prospective and (regarding study medication Acamprosate vs. Placebo) double blind design. A total of 371 patients has been randomly assigned immediately after detoxification to one of three different outpatient treat-ment conditions.

DETAILED DESCRIPTION:
The objective of this multi-center study is to optimize the long-term treatment of patients with alcohol dependence. This investigation should contribute to the issue of effective relapse prevention. Each treatment condition is lasting 6 months: a) Behavior Group Therapy + Acamprosate, b) Behavior Group Therapy + Placebo and c) support and counseling + Acamprosate. Follow-up examinations carried out 3 and 6 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSMIV criteria of alcoholism
* Age between 25 and 60
* Informed consent

Exclusion Criteria:

* Residence outside of the catchment area
* Legal reasons
* Insufficient knowledge of the German language
* Substance abuse or addiction other than alcohol or nicotine
* Pregnancy
* Serious physical illness
* Organic brain disease
* Contraindication to Acamprosate treatment

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 371 (Actual)
Dates: Start 2003-05; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Abstinence | 3,6,12 months

SECONDARY OUTCOMES:
Social functioning | 12 months
Cognitive functioning | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Gaebel, Professor, Study Chair — Department of Psychiatry and Psychotherapy, University of Düsseldorf
Locations (1):
- Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University Düsseldorf, Rhineland State Clinics Düsseldorf, Bergische Landstraße 2, 40629 Düsseldorf, Germany, Düsseldorf, North Rhine-Westfalia, Germany